CLINICAL TRIAL: NCT03318120
Title: Exercise Training in Dystonia and Other Involuntary Movement Disorders
Brief Title: Exercise Training in Dystonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201702224; 40115065 (Other: State of Florida); OCR28822 (Other: UF Oncore)
Record Dates: First submitted 2017-09-28; First posted 2017-10-23 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Dystonia
MeSH Terms: conditions — Dystonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Resistance Training (Experimental): Participants assigned to this arm will receive progressive resistance training under the supervision of a personal trainer at a gym facility close to their home. They will be required to perform these exercises twice a week for the first six months. They will be monitored with an activity monitor.
  Interventions: Behavioral: Progressive Resistance Training
- Control Arm (No Intervention): The control arm offered to subjects with dystonia and other involuntary muscle disorders, participants will be followed at baseline and 6 months similar to what will be done in active exercise arm but this arm will not receive exercise. They will be monitored with an activity monitor.

INTERVENTIONS:
Behavioral: Progressive Resistance Training — Participants will perform required resistance training exercises at regular intervals for a period of up to 3 years. They will be tested at a baseline visit, then every 6 months for a total of at least 5 visits. During these visits, they will be asked to complete the following: questionnaires about quality of life and depression, tests to measure strength and motor function, tests to measure cognition, an orientation session to learn a precision griping task, structural and functional MRI scans of the brain, measurement of brain waves using a non-invasive technique called electroencephalography (EEG) and muscle activity using electromyography (EMG), measurement of brain function with TMS, pregnancy test (if applicable).
  Arms: Progressive Resistance Training

SUMMARY:
The purpose of this research study is to investigate how the brain and motor behavior changes in individuals with dystonia and other involuntary movement disorders and healthy individuals over time with exercise training.

DETAILED DESCRIPTION:
The study team plan to conduct a randomized prospective, parallel-group, controlled study to examine the effects of exercises in dystonia and other involuntary movement disorders. Patients will be randomized to receive either progressive resistance training or a control treatment following the modified fitness protocol. The study team hypothesize that progressive resistance training will result in better outcomes compared to modified fitness protocol.

Data collect includes 1) data about clinical movement disorder history, age, gender, height, weight, and other medical conditions; 2) clinical neurological examination; 3) tests assessing cognitive abilities (the Montreal Cognitive Assessment, Stroop, Digit Span, Hopkins Verbal Learning Test, COWA and Animals, and Brief Test of Attention); 4) tests assessing motor abilities including Toronto Western Spasmodic Rating Scale (TWSTRS) and Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS); 5) measures of anxiety and depression (Beck Depression Index, Hamilton Anxiety and Depression Rating Scales); 5) Cervical dystonia related quality of life (CDQ-24); 6) Visual Analog Scales-Quality of Life (VAS QOL) evaluating of health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

Patients with dystonia and other involuntary movement disorders will be recruited whose diagnosis will be confirmed by a Movement Disorders specialist following the criteria recommended by movement disorders society.

* Patients will be eligible if they are ages 30 to 80 years,
* Receive stable doses of regular botulinum toxin injections and are on stable doses of oral pharmacological therapy if applicable, and are able to walk for 6 minutes.
* Age-matched healthy individuals will be recruited for normative data.
* All individuals must be capable of providing informed consent and complying with the study related procedures.

Exclusion Criteria:

Patients will be ineligible if they have a neurological history other than dystonia, have significant arthritis

* Fail the Physical Activity Readiness Questionnaire, have cognitive impairment as indicated by a Mini Mental State Examination score <23,
* Already exercising.
* As necessitated by the risks of Magnetic Resonance Imaging (MRI) or transcranial magnetic stimulation (TMS), patients who have any type of implanted electrical device (such as a cardiac pacemaker or a neurostimulator), or a certain type of metallic clip in their body (i.e., an aneurysm clip in the brain)
* Active seizure disorder are not eligible for participation in the MRI or TMS portion of the study.
* Individuals who are claustrophobic will also be excluded from participation.
* Women who are or might be pregnant and nursing mothers are not eligible. Pregnancy tests will be carried out for each female subject of child bearing potential prior to the participation in the study and prior to each follow up visit.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Toronto Western Spasmodic Torticollis Rating Scale Score | Baseline through 24 months
  Investigate changes in clinical function before and after exercise intervention. A 35 point clinical tool for assessing and documenting the status of patients with spasmodic torticollis (cervical dystonia).
Burke-Fahn-Marsden Dystonia Rating Scale score | Baseline through 24 months
  Investigate changes in clinical function before and after exercise intervention. This is a specific questionnaire for dystonia developed to assess the severity of the effect of dystonia on various parts of the body (eyes, mouth, speech/swallowing, neck, trunk, upper limb, and lower limb). Severity factors and provoking factors are rated on a scale from 0-4 and a total score is calculated.

SECONDARY OUTCOMES:
Transcranial Magnetic Stimulation (TMS) | Baseline through 24 months
  Investigate changes in motor cortex excitability via transcranial magnetic stimulation before and after exercise intervention
Oral Medication | Baseline through 24 months
  Investigate changes in oral medications taken by participants before and after exercise intervention
Changes in blood oxygen level-dependent (BOLD) signal | Baseline through 24 months
  Investigate changes in motor cortex excitability via blood oxygen level-dependent (BOLD) signal before and after exercise intervention
Hand grip dynamometer | Baseline through 24 months
  Investigate changes in maximum hand grip strength

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Wagle Shukla, M.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available without any personal identifiers included.